CLINICAL TRIAL: NCT05683756
Title: Optimizing Attention and Sleep Intervention Study: A Pilot RCT to Compare Parent Behavioral Interventions With and Without Sleep Strategies Delivered in Pediatric Primary Care for Preschool-aged Children at Risk of Childhood ADHD
Brief Title: Optimizing Attention and Sleep Intervention Study
Acronym: OASIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Heather Joseph, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22070096; R34MH131993 (NIH)
Record Dates: First submitted 2022-11-24; First posted 2023-01-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Hyperactivity Disorder; Child, Preschool; Sleep; Sleep Disturbance
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Attention Deficit Disorder with Hyperactivity; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Parent Behavioral Intervention (Active Comparator): A brief parent behavioral intervention with evidenced based strategies for treatment of ADHD.
  Interventions: Behavioral: Brief Parent Behavioral Intervention
- Sleep-Focused Parent Behavioral Intervention (Experimental): A modified version of the brief parent behavioral intervention that specifically targets sleep disrupting behaviors.
  Interventions: Behavioral: Sleep-Focused Parent Behavioral Intervention

INTERVENTIONS:
Behavioral: Brief Parent Behavioral Intervention — PBI administered in pediatric primary care by an embedded therapist.
  Arms: Brief Parent Behavioral Intervention
Behavioral: Sleep-Focused Parent Behavioral Intervention — SF-PBI administered in pediatric primary care by an embedded therapist.
  Arms: Sleep-Focused Parent Behavioral Intervention

SUMMARY:
The goal of this pilot clinical effectiveness trial is to compare a brief parent behavioral intervention (PBI) to a modified sleep focused PBI (SF-PBI) delivered by therapists in pediatric primary care for families of children 3-5 years old with sleep problems and early ADHD symptoms.

The main aims are to:

Aim 1: Demonstrate the acceptability, feasibility, and appropriateness of the sleep focused PBI (SF-PBI) delivered in pediatric primary care for preschool-aged children (3-5 years old) at elevated risk for ADHD.

Aim 2: Examine change in target engagement (sleep) and ADHD symptoms among preschool-aged children at elevated risk for ADHD receiving SF-PBI compared to standard PBI.

DETAILED DESCRIPTION:
Sleep problems may be one mechanism through which young children may be at risk for developing ADHD, although first line ADHD interventions, including parent behavioral interventions (PBIs), do not address sleep. Investigators will test a modified version of a PBI to target sleep disrupting behaviors for children 3-5 years old at elevated risk for ADHD. The intervention will be delivered by behavioral health therapists embedded in pediatric primary care to increase families' access to intervention. This pilot effectiveness trial is the first step towards developing an early intervention targeting sleep as a mechanism to reduce the prevalence, symptoms, and impairments associated with childhood ADHD.

ELIGIBILITY:
Inclusion Criteria:

Parent/Caregiver:

* (1) Legal guardian is at least 18 years of age
* (2) Reads and speaks English

Child:

* (1) 3-5 years of age
* (2) Caregiver report of 4 or more ADHD symptoms
* (3) Caregiver reports child's sleep as a "moderate" or "serious problem"
* (4) English speaking
* (5) Child receives care from participating pediatric primary care office

Exclusion Criteria:

* (1) Sleep interfering medical diagnoses (e.g., narcolepsy, obstructive sleep apnea)
* (2) Severe neurodevelopmental disorder

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability | Post Intervention at approximately 4 months
  Therapists and caregiver report of intervention acceptability will be assessed using the 4-item Acceptability of Intervention Measure (AIM), rated from 1-completely disagree to 5-completely agree, with scores greater than or equal to 16 indicating good acceptability.
Intervention Appropriateness | Post Intervention at approximately 4 months
  Therapists and caregiver report of intervention appropriateness will be assessed using the 4-item Intervention Appropriateness Measure (IAM), rated from 1-completely disagree to 5-completely agree, with scores greater than or equal to 16 indicating good appropriateness.
Intervention Feasibility | Post Intervention at approximately 4 months
  Therapists and caregiver report of intervention feasibility will be assessed using the 4-item Feasibility of Intervention Measure (FIM), rated from 1-completely disagree to 5-completely agree, with scores greater than or equal to 16 indicating good feasibility.
Problematic Sleep | Change from baseline up to 8 months
  Using the Brief Child Sleep Questionnaire caregivers will report on their perception of child's sleep as problematic, rated 1 (Not at all) to 5 (A serious problem).
ADHD Symptoms | Change from baseline up to 8 months
  Using the 18-item ADHD Rating Scale-IV-Preschool Version caregivers will report on the child's ADHD symptoms. Symptoms are rated from 0 (Rarely) to 3 (Very Often).

SECONDARY OUTCOMES:
Nighttime Awakenings | Change from baseline up to 8 months
  Caregivers will report how many times their child typically wakes during the night, using the Brief Child Sleep Questionnaire.
Sleep Latency | Change from baseline up to 8 months
  Sleep latency will be determined by using the caregiver report of how long it typically takes their child to fall asleep (number of minutes), using the Brief Child Sleep Questionnaire.
Consistency of Bedtime Routine | Change from baseline up to 8 months
  Caregivers will report the number of days, in a typical week, they regularly put their child to bed at the same time (within 15 minutes), using the Brief Child Sleep Questionnaire.

OTHER OUTCOMES:
Actigraphy | Change from baseline up to 8 months
  Actigraphy is collected for 10 days at each of the three study timepoints. These data are to assess feasibility of actigraphy data collection with this population and will be used in exploratory analyses.
Sleep Diary | Change from baseline up to 8 months
  Sleep diary is collected for 10 days at each of the three study timepoints. These data are to assess feasibility of parent reported sleep diary data collection with this population and will be used in exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Joseph, DO, Principal Investigator — Assistant Professor of Psychiatry and Pediatrics, University of Pittsburgh
Locations (7):
- United States (7):
  - Children's Community Pediatrics Bass Wolfson, Cranberry, Cranberry Township, Pennsylvania
  - Children's Community Pediatrics GIL Murrysville, Monroeville, Pennsylvania
  - Children's Community Pediatrics Shenango, New Castle, Pennsylvania
  - Children's Community Pediatrics Neshannock, New Castle, Pennsylvania
  - Children's Community Pediatrics GIL East Liberty, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Community Pediatrics Bass Wolfson, Squirrel Hill, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be shared, after deidentification, via the NIMH National Data Archive.
Supporting Information: Study Protocol
Time Frame: Data will be shared upon publication or 1 year after the grant end date. Data will be available indefinitely.
Access Criteria: Any NIMH NDA authorized users may request the data.
URL: https://nda.nih.gov

REFERENCES:
- [Background] Cunningham CE, Bremner R, Boyle M. Large group community-based parenting programs for families of preschoolers at risk for disruptive behaviour disorders: utilization, cost effectiveness, and outcome. J Child Psychol Psychiatry. 1995 Oct;36(7):1141-59. doi: 10.1111/j.1469-7610.1995.tb01362.x. PMID 8847377
- [Result] Joseph HM, Levenson JC, Conlon RPK, Mannion K, Kipp HL, Gradian A, Wallace ML, Williamson AA. Optimizing Attention and Sleep Intervention Study (OASIS): a protocol for a pilot randomized controlled trial to compare parent behavioral interventions with and without sleep strategies delivered in pediatric primary care for preschool-aged children at risk of childhood ADHD. Pilot Feasibility Stud. 2025 Feb 25;11(1):22. doi: 10.1186/s40814-025-01600-0. PMID 40001155